CLINICAL TRIAL: NCT07054151
Title: Clinical Predictors of Capillary Refill Time and Their Association With Triage Categories From the Emergency Department Perspective: A Cross-Sectional Study
Brief Title: Clinical Predictors of Capillary Refill Time and Their Association With Triage Categories
Acronym: CRT_TriageER
Status: Completed | Type: Observational
Sponsor: Izmir Democracy University (Other)
Responsible Party: Principal Investigator, Zeynep Sofuoglu, Assoc. Prof., Izmir Democracy University
Other Study IDs: IzmirDemocracy
Record Dates: First submitted 2025-05-21; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Triage; Emergency Medical Services; Vital Signs Monitoring; Hypoperfusion; Hemodynamic Instability
Keywords: Vital parameters; capillary refill time; prediction; Non-trauma Emergency; Emergency Medical Services; Triage; clinical decision-making

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non-traumatic patients admitted to the emergency department of Izmir Democracy University Buca Seyfi
  Interventions: Other: No clinical intervention (observational study only)

INTERVENTIONS:
Other: No clinical intervention (observational study only) — This is an observational study. No experimental or clinical intervention was applied. Only non-invasive data collection such as capillary refill time and vital sign measurements was performed.

SUMMARY:
This observational study aims to determine the correlation between capillary refill time (CRT) and vital parameters in patients presenting to the emergency department.

It explores whether CRT is associated with triage categories and vital signs in non-traumatic patients, including oxygen saturation (SpO₂), heart rate, systolic and diastolic blood pressure, body temperature, forearm temperature, and respiratory rate.

Patients admitted to the emergency department of a training and research hospital were assigned triage codes (green, yellow, red). Their CRT was measured three times, and vital signs were recorded accordingly.

DETAILED DESCRIPTION:
In the initial evaluation, patients admitted to the emergency department were assigned a triage color code, categorized as green, yellow, or red. In the color-coding system employed, green was designated as low urgency, yellow as medium urgency, and red as urgent. The allocation of triage codes is the responsibility of nurses who have undergone the requisite training. Following the completion of the assigned task, the emergency specialist proceeded to meticulously record a series of physiological parameters. These parameters included the CRT (in seconds), the percentage of oxygen saturation in the blood (SpO2%), the heart rate (in minutes), the systolic and diastolic blood pressure (in mmHg), the body temperature (in degrees Celsius), the forearm temperature measured at the CRT, and the respiratory rate (in minutes). CRT was evaluated three times for each patient, and the mean of these values was recorded as the CRT.

ELIGIBILITY:
Inclusion Criteria:

* individuals over the age of 18 years who consented to participate in the study

Exclusion Criteria:

* The presence of pregnancy
* Multiple traumas resulting in hypovolemia
* The absence of fingers or limbs
* The utilization of vasopressors or inotropic pharmacological agents
* The existence of peripheral arterial disease
* The presence of nail polish or fake nails

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of non-trauma patients who applied to the emergency department of Buca Research and Training Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 313 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Triage Code Assignment | Baseline [within 30 minutes of initial Emergency department admission triage assessment]
  Triage code assignment will be completed within the first 30 minutes of the patient's initial presentation to the emergency department (ED). Patients will be categorized into green, yellow, or red triage groups based on standard emergency triage protocols upon admission.
  Following this, the patient will be transferred to the designated emergency care room (ER) based on the assigned triage code and further clinical evaluation and treatment.
  Initially, the triage nurse will assess the patient and assign the triage code. Following this, the patient will be transferred to the designated emergency care room (ER), where a specialist emergency physician will perform further clinical evaluation and treatment.
Capillary Refill Time (CRT) in Seconds | Single measurement by the emergency physician within 10 minutes of the patient's arrival in the emergency care room
  CRT will be measured in seconds using a stopwatch after pressing the fingertip. The measurement will be repeated three times and average was calculated.Triage code assignment will be completed within the first 30 minutes of the patient's initial presentation to the emergency department (ED). Following this, the patient will be transferred to the designated emergency care room (ER) based on the assigned triage code, and all vital parameters (e.g., capillary refill time, heart rate, blood pressure) will be measured within 10 minutes of entering the emergency care area.
Heart Rate | The patient is then assessed by the emergency physician within 10 minutes of being transferred to the ER triage code section. (Single measurement )
  Heart rate will be recorded using standard clinical devices. Unit: Beats per minute Measurement technique:: Measured using clinical monitor.. Upon the patient's initial presentation to the emergency department (ED), triage code assignment will be completed within the first 30 minutes. Based on the assigned code, the patient will be directed to the appropriate emergency care room (ER). Heart rate measurements will be taken within 10 minutes of the patient's arrival in the emergency care room.
Systolic Blood Pressure | Single simultaneous measurement (systolic and diastolic) by the emergency physician within 10 minutes of arrival in the emergency care room (ER).
  systolic blood pressure will be recorded using standard clinical devices. Unit: mmHg Measurement technique: Measured using clinical monitor.
  Upon the patient's initial presentation to the emergency department (ED), triage code assignment will be completed within the first 30 minutes. Based on the assigned triage code, the patient will be directed to the appropriate emergency care room (ER).
  Systolic blood pressure will be measured once, within 10 minutes of the patient's arrival in the emergency care room.
  Systolic and diastolic blood pressure will be measured simultaneously in a single session within 10 minutes of the patient's arrival in the emergency care room.
Diastolic Blood Pressure | Single simultaneous measurement (systolic and diastolic) by the emergency physician within 10 minutes of arrival in the emergency care room (ER).
  diastolic blood pressure will be recorded using standard clinical devices. Unit: mmHg Measurement technique: Measured using clinical monitor. Upon the patient's initial presentation to the emergency department (ED), triage code assignment will be completed within 30 minutes. Based on the assigned triage code, the patient will be transferred to the appropriate emergency care room (ER).
  Diastolic and systolic blood pressure will be measured simultaneously in a single session within 10 minutes of the patient's arrival in the emergency care room.
SpO2 (Oxygen Saturation) | Single measurement by the emergency physician within 10 minutes of the patient's arrival in the emergency care room
  SpO2 will be recorded using standard clinical devices. Unit: Percent (%) Measurement technique: Measured using pulse oximetry. Oxygen saturation (SpO₂), along with other vital signs (blood pressure, heart rate), will be measured in a single session within 10 minutes of the patient's arrival in the emergency care room.
Respiratory Rate | Following the patient's admission to the ER, the triage nurse determins the patient's triage code. The patient is then assessed by the emergency physician within 10 minutes of being transferred to the ER triage code section. (single timepoint)
  respiratory rate will be recorded using standard clinical devices. Unit: Breaths per minute Measurement technique: Measured using observation and counting.
Forearm Temperature | Single measurement by the emergency physician within 10 minutes of the patient's arrival in the emergency care room (ER).
  Forearm temperature will be recorded using standard clinical devices. Unit: Degrees Celsius Measurement technique: Measured using infrared thermometer.
Body Temperature | Single measurement by the emergency physician within 10 minutes of the patient's arrival in the emergency care room (ER).
  Body temperature will be recorded using standard clinical devices. Unit: Degrees Celsius. Body temperature was measured with a Yobekan model KV-11 infrared measuring device.
  Measurement technique: Measured using infrared thermometer. All vital signs, including body temperature, were assessed sequentially by the same emergency physician within 10 minutes after the patient was transferred to the emergency care room (ER).

SECONDARY OUTCOMES:
Correlation Between Capillary Refill Time and Age | During the study period through data collection and data entry, expected to be completed within an average of 3 months.
  Pearson correlation analysis will be used to assess the correlation between capillary refill time (measured in seconds using a stopwatch and averaged from three measurements) and patient age (recorded in years from patient records).
  Unit of Measure:
  Capillary Refill Time (Mean): seconds Age: years
  Measurement Tool:
  CRT measured with a stopwatch by a trained emergency specialist Age extracted from patient record All CRT measurements will be taken within 10 minutes of the patient's arrival in the emergency care room by the same emergency physician, as part of the initial clinical evaluation.
Association Between Prolonged CRT (>2s) and Triage Category | During the study period through data collection and data entry, expected to be completed within an average of 3 months.
  Logistic regression will be used to assess the association between prolonged CRT (defined as >2 seconds, averaged from three measurements using a stopwatch) and triage category (Green, Yellow, Red) assigned at emergency department admission.
  Unit of Measure:
  CRT: seconds Triage: categorical (Green, Yellow, Red)
  Measurement Tool:
  CRT measured with a stopwatch (three repetitions, averaged) Triage assignment performed by certified triage nurse based on hospital protocol All CRT measurements were performed within 10 minutes of the patient's arrival in the emergency care room by the same emergency physician, as part of the initial vital sign assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Aysel Başer, Assoc.Prof., Study Director — Izmir Democracy University, Medical Faculty
Locations (1):
- Buca Training and Research Hospital, Emergency Deaprtment, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be shared with other researchers upon reasonable request, provided they submit a clear and justified explanation of their research purpose.
Supporting Information: ICF, Analytic Code
Time Frame: IPD and supporting document can be available between 01 September 2025 - 31 August 2028
Access Criteria: Access to the IPD will be granted to qualified researchers affiliated with academic or research institutions, upon submitting a research proposal that is approved by an independent ethics committee
URL: https://zenodo.org/records/15481027

REFERENCES:
- [Background] Adhikari S. Available at: www.jgpeman.com, eISSN: 2363-1168 28 SHORT REVIEW: CAPILLARY REFILLL VS SERUM LACTATE IN SEPTIC. Vol. 7, SHOCK Journal of General Practice and Emergency Medicine of Nepal. 2018.
- [Background] Sheridan DC, Kohn-Loncarica GA, Nunez P, Hudson R, Lin A, Samatham R, Hansen ML. Point-of-Care Noninvasive Technology for Pediatric Dehydration Assessment. Pediatr Emerg Care. 2023 Aug 1;39(8):569-573. doi: 10.1097/PEC.0000000000002824. Epub 2022 Oct 10. PMID 36252055
- [Background] Baker AH, Mazandi VM, Norton JS, Melendez E. Emergency Department Sepsis Triage Scoring Tool Elements Associated With Hypotension Within 24 Hours in Children With Fever and Tachycardia. Pediatr Emerg Care. 2024 Sep 1;40(9):644-649. doi: 10.1097/PEC.0000000000003153. Epub 2024 Mar 13. PMID 38471759
- [Background] Sheridan DC, Cloutier R, Kibler A, Hansen ML. Cutting-Edge Technology for Rapid Bedside Assessment of Capillary Refill Time for Early Diagnosis and Resuscitation of Sepsis. Front Med (Lausanne). 2020 Dec 21;7:612303. doi: 10.3389/fmed.2020.612303. eCollection 2020. PMID 33425956
- [Background] Jacquet-Lagreze M, Bouhamri N, Portran P, Schweizer R, Baudin F, Lilot M, Fornier W, Fellahi JL. Capillary refill time variation induced by passive leg raising predicts capillary refill time response to volume expansion. Crit Care. 2019 Aug 16;23(1):281. doi: 10.1186/s13054-019-2560-0. PMID 31420052
- [Background] Ait-Oufella H, Bige N, Boelle PY, Pichereau C, Alves M, Bertinchamp R, Baudel JL, Galbois A, Maury E, Guidet B. Capillary refill time exploration during septic shock. Intensive Care Med. 2014 Jul;40(7):958-64. doi: 10.1007/s00134-014-3326-4. Epub 2014 May 9. PMID 24811942
- [Background] Faul A, Lang. Correlation Problems Referring to One Correlation Comparison of a correlation with a constant 0 (bivariate normal model) Comparison of a correlation with 0 (point biserial model) Comparison of a correlation with a constant 0 (tetrachoric correlation model).
- [Background] Sansone CM, Prendin F, Giordano G, Casati P, Destrebecq A, Terzoni S. Relationship between Capillary Refill Time at Triage and Abnormal Clinical Condition: A Prospective Study. Open Nurs J. 2017 Jul 26;11:84-90. doi: 10.2174/1874434601711010084. eCollection 2017. PMID 28839512
- [Background] Schriger DL, Baraff L. Defining normal capillary refill: variation with age, sex, and temperature. Ann Emerg Med. 1988 Sep;17(9):932-5. doi: 10.1016/s0196-0644(88)80675-9. PMID 3415066
- [Background] Jacquet-Lagreze M, Wiart C, Schweizer R, Didier L, Ruste M, Coutrot M, Legrand M, Baudin F, Javouhey E, Depret F, Fellahi JL. Capillary refill time for the management of acute circulatory failure: a survey among pediatric and adult intensivists. BMC Emerg Med. 2022 Jul 18;22(1):131. doi: 10.1186/s12873-022-00681-x. PMID 35850662
- [Background] Lewin J, Maconochie I. Capillary refill time in adults. Emerg Med J. 2008 Jun;25(6):325-6. doi: 10.1136/emj.2007.055244. No abstract available. PMID 18499809
- [Background] Hazinski MF, Zaritsky AL, Nadkarni CD. PALS Provider Manual. Dallas: American Heart Association; 2002.
- [Background] Van der Mullen J, Wise R, Vermeulen G, Moonen PJ, Malbrain MLNG. Assessment of hypovolaemia in the critically ill. Anaesthesiol Intensive Ther. 2018;50(2):141-149. doi: 10.5603/AIT.a2017.0077. Epub 2017 Nov 28. PMID 29182211
- [Background] McGuire D, Gotlib A, King J. Capillary Refill Time. 2023 Apr 23. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK557753/ PMID 32491685
- [Background] Champion HR, Sacco WJ, Hannan DS, Lepper RL, Atzinger ES, Copes WS, Prall RH. Assessment of injury severity: the triage index. Crit Care Med. 1980 Apr;8(4):201-8. doi: 10.1097/00003246-198004000-00001. PMID 7357873
- [Background] Champion HR, Sacco WJ, Carnazzo AJ, Copes W, Fouty WJ. Trauma score. Crit Care Med. 1981 Sep;9(9):672-6. doi: 10.1097/00003246-198109000-00015. PMID 7273818
- [Background] BEECHER HK, SIMEONE FA, et al. The internal state of the severely wounded man on entry to the most forward hospital. Surgery. 1947 Oct;22(4):672-711. No abstract available. PMID 20266131
- [Background] Pickard A, Karlen W, Ansermino JM. Capillary refill time: is it still a useful clinical sign? Anesth Analg. 2011 Jul;113(1):120-3. doi: 10.1213/ANE.0b013e31821569f9. Epub 2011 Apr 25. PMID 21519051
- See also: DataSet — https://zenodo.org/records/15481027